CLINICAL TRIAL: NCT04853121
Title: Accuracy and Primary Stability of Straight and Tapered Implants Placed Into Fresh Extraction Sockets Using Dynamic Navigation
Brief Title: Accuracy and Primary Stability of Straight and Tapered Implants in Immediate Implant Placement Using Dynamic Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Junyu Shi, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SH9H-2020-T410-2
Record Dates: First submitted 2021-03-23; First posted 2021-04-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Tooth Diseases
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tapered implant (Active Comparator)
  Interventions: Procedure: Tapered Implants
- straight implant (Placebo Comparator)
  Interventions: Procedure: Straight Implants

INTERVENTIONS:
Procedure: Tapered Implants — Tapered Implants are placed in fresh socket via dynamic navigation
  Arms: tapered implant
Procedure: Straight Implants — Straight Implants are placed in fresh socket via dynamic navigation
  Arms: straight implant

SUMMARY:
Prosthetic-driven immediate implant placement for optimal aesthetic restoration has been increasing in demand during the last decades but requires higher accuracy. Dynamic navigation has been a reported better implant positioning. There are two main choices of implant macrogeometry: straight and tapered implants. One feature of implant design that may influence implants' accuracy is the taper of the implant body. However, their exact role is still needed to be investigated further. Besides, implant macrogeometry may influence primary stability, which is a prerequisite in achieving osseointegration. Therefore, we designed a randomized controlled clinical trial study to verify the clinical efficacy of the implant macrogeometry by comparing straight implants with tapered implants in immediate implant placement using dynamic navigation.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and in good health;
2. The maxillary incisor that cannot be retained due to non-periodontitis;
3. The buccal bone plate is complete;
4. No acute infection;
5. The extraction socket have at least 3-5 mm apical bone.

Exclusion Criteria:

1. General contraindications of oral implant surgery (such as immunodeficiency, long-term use of corticosteroids);
2. Treatments or diseases that may affect bone tissue metabolism (for example, taking bisphosphonates or receiving local radiotherapy);
3. Periodontitis history or uncontrolled periodontitis. Bleeding of probing (BOP) positive site ≥ 10%, or probing depth (PD) ≥ 4mm;
4. Heavy smokers or previous heavy smoking history (quit smoking time <5 years or> 20 cigarettes per day);
5. Refuse to participate in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Accuracy | one week
  mm

SECONDARY OUTCOMES:
Insetion torque value, ITV | surgery day
  to detect primary stability
Implant Stability Quotient, ISQ | surgery day
  to detect primary stability

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China